CLINICAL TRIAL: NCT05307757
Title: Diffusion-Weighted MRI for Screening Contralateral Breast Cancers in Patients With Newly Diagnosed Breast Cancer
Brief Title: Screening Contralateral Breast Cancers in Patients With Newly Diagnosed Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: Contralateral Screening
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In women with newly diagnosed breast cancer, synchronous contralateral breast cancer is reported in 1% to 3%. During the initial diagnosis of breast cancer, it is important to detect the contralateral cancer to avoid second round of cancer therapy. Because breast MRI is a highly sensitive modality, it is used for screening of occult contralateral disease in women newly diagnosed with breast cancer and detects contralateral cancers not seen on clinical or conventional imaging (mammography and ultrasonography) in 4.1% of women. However, the use of breast MRI for screening contralateral breast cancer, is limited not only by high costs and long examination time but also by high false-positive findings resulting in more benign biopsies and extensive surgeries. In addition, the use of intravenous gadolinium-based contrast agent is contraindicated in pregnancy and in women with renal impairment or contrast material allergy contrast. Thus, there is a need to develop a more safe and cost-effective supplemental imaging modality for screening breast cancer. Diffusion-weighted (DW) MRI is a fast, functional modality that measures the movement of water molecules to create tissue contrast without the need for contrast injection. Breast malignancies exhibit hindered diffusion and appear hyperintense on DW MRI with low apparent diffusion coefficient (ADC) compared to normal surrounding tissue. A number of studies have shown that the use of DW MRI can significantly reduce the false positives and unnecessary benign biopsy of breast MRI. Several studies have explored how to use DW MRI as a stand-alone tool for breast cancer screening, and recent results have shown that DW MRI is more useful than conventional imaging in detecting small breast cancer. However, most of these studies were retrospective with inconsistent results. Thus, a prospective multicenter study with standardized acquisition and interpretation protocols in a large population is needed to determine the efficacy of DW MRI for breast cancer screening. The purpose of our study is to determine whether DWI improves the performance of preoperative DCE MRI in detecting clinically occult contralateral breast cancers.

DETAILED DESCRIPTION:
* This is a multicenter, intraindividual comparative cohort study.
* A total of 1098 women with newly diagnosed breast cancer will be enrolled in this study.
* Each eligible woman with newly diagnosed invasive breast cancer will undergo DCE MRI and DWI at a 3T MR scanner.
* Contrast-enhanced MRI and DWI will be interpreted independently according to the Breast Imaging Reporting and Data System (BI-RADS) and likelihood of malignancy (Score range, 0%-100%) by trained radiologists.
* BI-RADS final assessment score of 3, 4 or 5 are considered to be positive.
* Pathology of core or surgical biopsy and 2 year follow up is the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Women aged more than 25 years at the time of enrollment
* Women underwent digital mammography and whole-breast US before MRI
* Women with image-guided biopsy result of invasive breast cancer
* Women who are planning for breast conservation surgery
* Women who will undergo preoperative breast MRI

Exclusion Criteria:

1. Women aged less than 25 years at the time of enrollment
2. Women with image-guided biopsy result of ductal carcinoma in situ or recurrent breast cancer
3. Women who underwent lumpectomy before MRI
4. Women receiving neoadjuvant chemotherapy or undergoing chemotherapy due to other malignancy
5. Pregnant or lactating women
6. Women with contraindication to breast MRI (claustrophobia, renal insufficiency GFR <60mL/min/1.73m2, metallic foreign body, history of severe side effects due to MR contrast agent, who cannot tolerate 40 minute scanning time etc).

Ages: 25 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with Newly Diagnosed Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The area under the (receiver operating characteristic) curve (AUC) per lesion and breast level | 2 year after enrollment
  AUC

SECONDARY OUTCOMES:
Sensitivity per lesion and breast level | 2 year after enrollment
  Number of positive examinations with a tissue diagnosis of cancer within 2 year/All examinations with tissue diagnosis of cancer within the same period
Specificity per lesion and breast level | 2 year after enrollment
  Number of negative examinations without tissue diagnosis of cancer within 2 year/All examinations without tissue diagnosis of cancer within the same period
Positive Predictive value per lesion and breast level | 2 year after enrollment
  True positive/True positive + False positive
Characteristics of detected cancers | 2 year after enrollment
  Tumor size, type, grade, molecular subtype, and lymph node metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park VY, Shin HJ, Kang BJ, Kim MJ, Moon WK, Song SE, Ha SM. Diffusion-Weighted Magnetic Resonance Imaging for Preoperative Evaluation of Patients With Breast Cancer: Protocol of a Prospective, Multicenter, Observational Cohort Study. J Breast Cancer. 2023 Jun;26(3):292-301. doi: 10.4048/jbc.2023.26.e18. Epub 2023 Apr 6. PMID 37272245